CLINICAL TRIAL: NCT05242484
Title: A Phase 2b Randomized, Double-blind, Active-and Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Induction and Maintenance Combination Therapy With Guselkumab and Golimumab in Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Combination Therapy With Guselkumab and Golimumab in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: DUET-UC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109179; 78934804UCO2001 (Other: Janssen Research & Development, LLC); 2021-005528-39 (EudraCT Number); 2023-504743-13-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-02-15; First posted 2022-02-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — guselkumab; golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: Placebo (Placebo Comparator): Participants will receive placebo subcutaneously (SC). All participants who meet inadequate response criteria will be escalated to an active treatment. Participants who are eligible and willing to continue the study intervention that they are receiving at Week 44 may enter the long-term extension.
  Interventions: Drug: Placebo
- Group 2: Guselkumab (Experimental): Participants will receive guselkumab dose regimen 1 SC. All participants who meet inadequate response criteria will be escalated to an active treatment. Participants who are eligible and willing to continue the study intervention that they are receiving at Week 44 may enter the long-term extension.
  Interventions: Biological: Guselkumab
- Group 3: Golimumab (Experimental): Participants will receive golimumab dose regimen 1 SC. All participants who meet inadequate response criteria will be escalated to an active treatment. Participants who are eligible and willing to continue the study intervention that they are receiving at Week 44 may enter the long-term extension.
  Interventions: Biological: Golimumab
- Group 4: JNJ-78934804 (High-dose) (Experimental): Participants will receive JNJ-78934804 dose regimen 1 SC. All participants who meet inadequate response criteria will be escalated to an active treatment. Participants who are eligible and willing to continue the study intervention that they are receiving at Week 44 may enter the long-term extension.
  Interventions: Biological: JNJ-78934804
- Group 5: JNJ-78934804 (Mid-dose) (Experimental): Participants will receive JNJ-78934804 dose regimen 2 SC. All participants who meet inadequate response criteria will be escalated to an active treatment. Participants who are eligible and willing to continue the study intervention that they are receiving at Week 44 may enter the long-term extension.
  Interventions: Biological: JNJ-78934804
- Group 6: JNJ-78934804 (Low-dose) (Experimental): Participants will receive JNJ-78934804 dose regimen 3 SC. All participants who meet inadequate response criteria will be escalated to an active treatment. Participants who are eligible and willing to continue the study intervention that they are receiving at Week 44 may enter the long-term extension.
  Interventions: Biological: JNJ-78934804

INTERVENTIONS:
Biological: Guselkumab — Guselkumab will be administered as subcutaneous injection.
  Arms: Group 2: Guselkumab
Biological: Golimumab — Golimumab will be administered as subcutaneous injection.
  Arms: Group 3: Golimumab
Biological: JNJ-78934804 — JNJ-78934804 will be administered subcutaneously as per defined regimen.
  Arms: Group 4: JNJ-78934804 (High-dose); Group 5: JNJ-78934804 (Mid-dose); Group 6: JNJ-78934804 (Low-dose)
Drug: Placebo — Placebo will be administered as subcutaneous injection.
  Arms: Group 1: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of JNJ-78934804 as compared to guselkumab and golimumab in participants with moderately to severely active ulcerative colitis who have had an inadequate initial response, loss of response, or intolerance to one or more approved advanced therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ulcerative colitis (UC) for at least 3 months prior to baseline
* Moderately to severely active UC as assessed by the modified Mayo score
* Demonstrated inadequate response, loss of response, or intolerance to at least one biologic or novel oral with biologic-like activity
* If female and of childbearing potential, must meet the contraception and reproduction requirements

Exclusion Criteria:

* Has severe extensive colitis as defined in the protocol
* Extent of inflammatory disease limited to the rectum
* Participants with current diagnosis of indeterminate colitis, microscopic colitis, ischemic colitis, or Crohn's disease (CD)
* Has a history of, or ongoing, chronic or recurrent infectious disease, including but not limited to, sinopulmonary infections, bronchiectasis, recurrent renal/urinary tract infections (example, pyelonephritis, cystitis), an open, draining, or infected skin wound, or an ulcer
* Currently has a malignancy or a history of malignancy within 5 years before screening (with the exception of nonmelanoma skin cancer or cervical carcinoma in situ that has been treated with no evidence of recurrence within 12 months of first dose of study intervention)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2029-03-27 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 48 | Week 48
  Percentage of participants with clinical remission at Week 48 will be reported. Clinical remission based on the modified Mayo subscores.

SECONDARY OUTCOMES:
Percentage of Participants with Endoscopic Improvement at Week 48 | Week 48
  Percentage of participants with endoscopic improvement at Week 48 will be reported. Endoscopic improvement at Week 48 based on the Mayo endoscopic subscore.
Percentage of Participants with Corticosteroid-free Clinical Remission at Week 48 | Week 48
  Percentage of participants with corticosteroid-free (60-day) clinical remission at Week 48 will be reported.
Percentage of Participants with Symptomatic Remission at Week 48 | Week 48
  Percentage of participants with symptomatic remission at Week 48 will be reported. Symptomatic remission at Week 48 based on stool and rectal bleeding symptoms.
Percentage of Participants with Combination of Histological Remission and Endoscopic Improvement at Week 48 | Week 48
  Percentage of participants with combination of histological remission and endoscopic improvement at Week 48 will be reported. Histologic remission and endoscopic improvement at Week 48 based on the histologic grading and the Mayo endoscopy subscore.
Secondary Comparison: Percentage of Participants with Clinical Remission at Week 48 | Week 48
  Percentage of participants with clinical remission at Week 48 will be reported. Clinical remission based on the modified Mayo subscores will be reported.
Percentage of Participants with Adverse Events (AEs) | Up to Week 48
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Percentage of Participants with Serious Adverse Events (SAEs) | Up to Week 48
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Laboratory Parameters Over Time | Up to Week 48
  Laboratory parameters over time will be reported.
Vital Signs Parameters Over Time | Up to Week 48
  Vital signs parameters over time will be reported.
Suicidal Ideation Assessment Using Columbia Suicide Severity Rating Scale (C-SSRS) Score | Up to Week 48
  The C-SSRS scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Worsening of suicidal ideation was an increase in severity of suicidal ideation from baseline.
Serum Concentrations of Guselkumab Over Time | Up to Week 48
  Serum concentrations of guselkumab over time will be reported. Serum samples will be analyzed to determine concentrations of guselkumab using a validated, specific, and sensitive method.
Serum Concentrations of Golimumab Over Time | Up to Week 48
  Serum concentration of golimumab over time will be reported. Serum samples will be analyzed to determine concentrations of golimumab using a validated, specific, and sensitive method.
Percentage of Participants with Antibodies to Guselkumab | Up to Week 48
  Percentage of participants with antibodies to guselkumab will be reported.
Titers of Antibodies to Guselkumab | Up to Week 48
  Titers of antibodies to guselkumab will be reported.
Percentage of Participants with Antibodies to Golimumab | Up to Week 48
  Percentage of Participants with Antibodies to golimumab will be reported.
Titers of Antibodies to Golimumab | Up to Week 48
  Titers of antibodies to golimumab will be reported.
Percentage of Participants with Neutralizing Antibodies to Guselkumab | Up to Week 48
  Percentage of participants with neutralizing antibodies to guselkumab will be reported.
Percentage of Participants with Neutralizing Antibodies to Golimumab | Up to Week 48
  Percentage of participants with neutralizing antibodies to golimumab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (402):
- United States (63):
  - Valley Gastroenterology Medical Group, Arcadia, California
  - Southern California Research Center, Coronado, California
  - Om Research LLC, Lancaster, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Medical Research Center of Connecticut, Hamden, Connecticut
  - Yale University, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Pioneer Research Solutions Inc., Coconut Creek, Florida
  - Digestive and Liver Disease Institute, Kissimmee, Florida
  - Osceola Regional Hospital, Kissimmee, Florida
  - Florida Research Center Inc., Lakewood Rch, Florida
  - University of Miami, Miami, Florida
  - Gastroenterology Group Of Naples, Naples, Florida
  - Omega Research Consultants, Orlando, Florida
  - Synergy Clinical Research, St. Petersburg, Florida
  - GCP Clinical Research, Tampa, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastroenterolgy Associates of Central GA, Macon, Georgia
  - Atlanta Gastroenterology Associates, Marietta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Gastroenterology Consultants, Roswell, Georgia
  - Grand Teton Gastroenterology, Idaho Falls, Idaho
  - IU Health University Hospital, Indianapolis, Indiana
  - Gastroenterology of Southern Indiana, New Albany, Indiana
  - Tri-State Gastroenterology Assoc, Crestview Hills, Kentucky
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham And Women's Hospital, Chestnut Hill, Massachusetts
  - Huron Gastroenterology Associates Center for Digestive Care, Ypsilanti, Michigan
  - Washington University, St Louis, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Care Access Las Vegas, Las Vegas, Nevada
  - Dartmouth Hitchcock, Lebanon, New Hampshire
  - Weill Cornell Medical College, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Mohawk Valley Endoscopy Center, Utica, New York
  - University North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Tryon Medical Group, Charlotte, North Carolina
  - Onsite Clinical Solutions, Charlotte, North Carolina
  - Care Access Research, Kinston, Kinston, North Carolina
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Frontier Clinical Research, Uniontown, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Digestive Disease Associates, Rock Hill, South Carolina
  - Gastro One, Germantown, Tennessee
  - Etsu Quillen College Of Medicine, Johnson City, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - GI Specialists of Houston, Houston, Texas
  - Gastroenterology Clinic Of San Antonio P A, San Antonio, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Medical College Of Virginia Hospital, Richmond, Virginia
  - Washington Gastroenterology, PLLC, Bellevue, Washington
  - Swedish Medical Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Digestive Health Specialists, Tacoma, Washington
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Argentina (6):
  - CIPREC, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Hospital de Gastroenterología Dr. Carlos Bonorino Udaondo, Ciudad Autonoma Buenos Aires
  - Sanatorio Duarte Quiroz, Córdoba
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Hospital Provincial del Centenario, Rosario
- Australia (11):
  - Box Hill Hospital, Box Hill
  - Royal Prince Alfred Hospital, Camperdown
  - Monash Health, Monash Medical Centre, Clayton
  - Concord Hospital, Concord
  - Western Health, Footscray
  - Coastal Digestive Health, Maroochydore
  - Fiona Stanley Hospital, Murdoch
  - Royal Adelaide Hospital, North Terrace
  - Royal Melbourne Hospital, Parkville
  - The Alfred Hospital, Prahran
  - Mater Hospital Brisbane, South Brisbane
- Austria (4):
  - Universitaetsklinikum Salzburg Landeskrankenhaus, Salzburg
  - Krankenhaus der Barmherzigen Brüder, Vienna
  - Medizinische Universitaet Wien, Vienna
  - Klinikum Wels Grieskirchen, Wels
- Belgium (9):
  - Imelda Ziekenhuis, Bonheiden
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Cliniques Universitaires Saint Luc, Brussels
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHC MontLegia, Liège
  - CHU de Liege, Liège
  - Vitaz, Sint-Niklaas
- Brazil (16):
  - Universidade Estadual Paulista 'Julio De Mesquita Filho', Botucatu
  - L2IP Instituto de Pesquisas Clinicas, Brasília
  - Chronos Clinica Medica LTDA Chronos Pesquisa Clinica, Brasília
  - Fundacao Universidade de Caxias do Sul, Caxias do Sul
  - Centro Digestivo de Curitiba - Instituto de Pesquisa Clínica, Curitiba
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Hospital De Clinicas De Porto Alegre, Porto Alegre
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Universidade Federal do Rio de Janeiro - Faculdade de Medicina, Rio de Janeiro
  - SER - Servicos Especializados em Reumatologia da Bahia, Salvador
  - Pesquisare Saude, Santo André
  - Irmandade da Santa Casa da Misericórdia de Santos, Santos
  - Hospital Nove de Julho, São Paulo
  - BR Trials, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual IAMSPE, São Paulo
  - Instituto D Or de Pesquisa e Ensino IDOR, São Paulo
- Bulgaria (6):
  - Medical Centre Hipocrat, Haskovo
  - Diagnostic Consulting Center I Sliven, Sliven
  - UMHAT 'Tsaritsa Yoanna', Sofia
  - University Hospital Alexandrovska - Clinic of Nephrology, Sofia-Grad
  - Medical Center -Medika Plus, Veliko Tarnovo
  - Multriprofile Hospital for Active Treatment Hristo Botev, Vratsa
- Canada (19):
  - Foothills Hospital, Calgary, Alberta
  - Gastroenterology and Internal Medicine Research Institute (GIRI), Edmonton, Alberta
  - Covenant Health/Grey Nuns hospital, Edmonton, Alberta
  - Columbia Gastroenterology, New Westminster, British Columbia
  - The Gordon & Leslie Diamond Health Care Center, Vancouver, British Columbia
  - GIRI Gastrointestinal Research Institute, Vancouver, British Columbia
  - The Medical Arts Health Research Group, Vancouver, British Columbia
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - Viable Clinical Research, Dartmouth, Nova Scotia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - London Health Sciences Centre - University Campus, London, Ontario
  - Toronto Immune and Digestive Health Institute Inc, Toronto, Ontario
  - CIUSSS de l Est de l Ile de Montreal Installation Hopital Maisonneuve Rosemont, Montreal, Quebec
  - McGill University - Health Centre - Montreal General Hospital, Montreal, Quebec
  - CMIIM, Centre médical L'Enjeu, Mount Royal, Quebec
  - St. Jerome Medical Research, Saint-Jérôme, Quebec
  - Viable Clinical Research, Bridgewater
  - Hopital Chicoutimi, Saguenay
- Chile (4):
  - Hospital Clinico Regional Dr. Guillermo Grant Benavente, Concepción
  - Clinica Dermacross S A, Santiago
  - Complejo Asistencial Hospital Dr. Sótero del Río, Santiago
  - Centro de Estudios Clínicos e Investigación Médica (CeCim), Santiago
- China (6):
  - China Japan Friendship Hospital, Chaoyang
  - West China Hospital Sichuan University, Chengdu
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Jinhua municipal central hospital, Jinhua
  - Zhongda Hospital Southeast University, Nanjing
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
- Croatia (3):
  - Opca bolnica Bjelovar, Bjelovar
  - University Hospital Center Split, Split
  - University Hospital Dubrava, Zagreb
- Czechia (2):
  - Vojenska nemocnice Brno, Brno
  - ISCARE a.s., Prague
- Denmark (5):
  - Aalborg Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Bispebjerg Og Frederiksberg Hospital, Copenhagen
  - Herlev Hospital, University of Copenhagen, Herlev
  - Odense Universitetshospital, Odense
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- France (16):
  - CHU Amiens - Hopital Sud, Amiens
  - Hopital Louis Mourier, Colombes
  - Centre Hospitalier Universitaire(CHU) - Hopital Henri Mondor, Créteil
  - CHU Grenoble, Grenoble
  - Centre Hospitalier Départemental VENDEE, La Roche-sur-Yon
  - CHRU de Lille Hopital Claude Huriez, Lille
  - Hopital Nord Marseille, Marseille
  - Hopital Saint Eloi, Montpellier
  - Clinique Ambroise Pare, Neuilly-sur-Seine
  - CHU de Nice Hopital de l Archet, Nice
  - CHU Nimes Hopital Caremeau, Nîmes
  - Hopital Haut-Leveque, CMC Magellan, Pessac
  - Hospices Civils de Lyon HCL, Pierre-Bénite
  - CHU Saint Etienne, Saint-Etienne
  - Hopital de Rangueil, Toulouse
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy
- Germany (32):
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Praxis Fur Gastroenteroligie, Berlin
  - Charite - Universitaetsmedizin Berlin (CCM), Berlin
  - Krankenhaus Waldfriede Mitte, Berlin
  - University Hospital Dresden, Dresden
  - Universitaetsklinik Erlangen, Erlangen
  - JWG-University Hospital, Frankfurt
  - Agaplesion Frankfurter Diakonie Kliniken GmbH, Markus Krankenhaus, Frankfurt am Main
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Fulda - Tumorklinik - Germany, Fulda
  - Martin-Luther-Universitaet Halle-Wittenberg - Universitaetsk, Halle
  - BSF Studiengesellschaft, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Gastroenterology Outpatient Clinic Prof. Ehehalt/Dr. Hemstäd, Heidelberg
  - University Hospital Heidelberg, Heidelberg
  - Universitatsklinikum Jena, Jena
  - Praxisgemeinschaft Jerichow, Jerichow
  - Gastroenterologische Spezialpraxis - Berlin-Karlshorst, Karlshorst
  - Eugastro GmbH, Leipzig
  - Staedtisches Klinikum Lueneburg, Lüneburg
  - Universitaetsklinikum Mannheim, Mannheim
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Klinikum der Universitaet Muenchen, Munich
  - Praxis fur Innere Medizin und Gastroenterologie, Münster
  - MVZ Portal 10, Münster
  - Medius Klinik Nurtingen, Nürtingen
  - Siloah St Trudpert Klinikum, Pforzheim
  - Zentrum für Gastroenterologie Saar MVZ GmbH, Saarbrücken
  - Universitaetsklinik Tuebingen, Tübingen
  - Universitatsklinikum Ulm, Ulm
  - Gemeinschaftspraxis Jakobeit, Wipperfürth
  - Universitatsklinikum Wurzburg, Würzburg
- Greece (4):
  - Sotiria General State Hospital of Chest Diseases, Athens
  - Alexandra General Hospital of Athens, Athens
  - Nikaia General Hospital, Piraeus
  - Hippokration Hospital, Thessaloniki
- Hungary (7):
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis Egyetem, Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
  - Bugat Pal Korhaz, Gyöngyös
  - Szegedi Tud Egyetem Szent Gyorgyi Albert Klin Kozp, Szeged
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
- India (9):
  - M S Ramaiah Medical College and Hospital, Bangalore
  - Siksha O Anusandhan University - Institute of Medical Scienc, Bhubaneswar
  - Apex Hospitals Ltd, Jaipur
  - G.B. Pant Hospital, New Delhi
  - All India Institute of Medical Sciences, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Fortis Hospital, New Delhi
  - Yashoda Super Speciality Hospitals, Secunderabad
  - Surat Institute of Digestive Sciences Hospitals, Surat
- Israel (10):
  - Haemek Medical Center - Afula, Afula
  - Rambam Medical Center, Haifa
  - Bnai Zion Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Hebrew University Medical Center, Jerusalem
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Center, Tzrifin
- Italy (12):
  - Università degli Studi di Bari, Bari
  - A.O. Per L' Emergenza Cannizzaro - U.O. Chirurgia Generale, Catania
  - AOU Policlinico G.Martino, Messina
  - Ospedale San Raffaele HSR Istituto Scientifico Universitario San Raffaele, Milan
  - Azienda Ospedaliero Universitaria di Cagliari - Policlinico Duilio Casula di Monserrato, Monserrato
  - Azienda Ospedaliera San Gerardo, Monza
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - Ospedale Villa Sofia-Cervello, Palermo
  - Università Campus Biomedico di Roma, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - IRCCS Humanitas Rozzano-IBD Center Malattie Infiammatorie Croniche Intestinali, Rozzano
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Japan (52):
  - Asahikawa Medical University Hospital, Asahikawa
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Kitakyushu Municipal Medical Center, Fukuoka-ken
  - Gifu Prefectural General Medical Center, Gifu
  - Tokai University Hachioji Hospital, Hachiōji
  - Hamamatsu University Hospital, Hamamatsu
  - National Hospital Organization Hirosaki General Medical Center, Hirosaki
  - Hirosaki University Hospital, Hirosaki
  - Tokai University Hospital, Isehara
  - Kagoshima University Hospital, Kagoshima
  - Kagoshima IBD Gastroenterology Clinic, Kagoshima
  - Ofuna Chuo Hospital, Kamakura
  - Matsushima Clinic, Kanagawa
  - Nara Medical University Hospital, Kashihara
  - Tsujinaka Hospital Kashiwanoha, Kashiwa
  - Kobe University Hospital, Kobe
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kumamoto University Hospital, Kumamoto
  - Kurume University Hospital, Kurume
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University Hospital, Kyoto
  - Gunma University Hospital, Maebashi
  - Kitasato University Kitasato Institute Hospital, Minatoku
  - Kyorin University Hospital, Mitaka
  - Iwate Medical University Hospital, Morioka
  - Nagoya University Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - The Hospital of Hyogo College of Medicine, Nishinomiya
  - Kinshukai Infusion Clinic, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka City University Hospital, Osaka
  - Japan Community Health Care Organization Osaka Hospital, Osaka
  - Ogaki Municipal Hospital, Ōgaki
  - Oita Red Cross Hospital, Ōita
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Tokushukai Hospital, Sapporo
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Sapporo
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Sapporo IBD Clinic, Sapporo Chuo-ku
  - Tokyo Metropolitan Bokutoh Hospital, Sumida Ku
  - The Jikei University Hospital, Tokyo
  - Tokyo Saiseikai Central Hospital, Tokyo
  - National Hospital Organization Tokyo Medical Center, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Oji General Hospital, Tomakomai
  - Toyama Prefectural Central Hospital, Toyama
  - Toyota Kosei Hospital, Toyota
  - Mie University Hospital, Tsu
  - University of Tsukuba Hospital, Tsukuba
  - Wakayama Medical University Hospital, Wakayama
  - Yokohama City University Medical Center, Yokohama
- Jordan (4):
  - Istishari Hospital, Amman
  - Jordan University Hospital, Amman
  - Irbid Specialty Hospital, Irbid
  - King Abdullah University Hospital, Irbid
- Netherlands (5):
  - Academisch Medisch Centrum Universiteit van Amsterdam, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Maastricht University Medical Centre, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
  - UMC Utrecht, Utrecht
- New Zealand (4):
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Hutt Hospital, Lower Hutt
  - Wellington Hospital, Wellington
- Norway (6):
  - Alesund sjukehus, Ålesund
  - Vestre Viken HF Baerum Sykehus, Gjettum
  - Sykehuset Innlandet HF Gjøvik, Gjøvik
  - Akershus Universitetssykehus, Lørenskog
  - Oslo University Hospital HF Ulleval sykehus, Oslo
  - Universitetssykehuset Nord-Norge HF, Tromsø
- Poland (26):
  - Szpital Uniwersytecki No2, Bydgoszcz
  - Centrum Medyczne Plejady, Krakow
  - Centrum Medyczne Promed, Krakow
  - AmiCare Centrum Medyczne, Lodz
  - ETG Lublin, Lublin
  - Gastromed Spotka Z Ograniczona Odpowiedzialnoscia Sp. K., Lublin
  - Allmedica, Nowy Targ
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Synexus Polska Sp z o o, Poznan
  - Twoja Przychodnia, Poznan
  - Centrum Medyczne Medyk, Rzeszów
  - Endoskopia Sp z o.o., Sopot
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Sonomed Sp. z o.o., Szczecin
  - GASTROMED Sp. z o.o., Torun
  - Centrum Zdrowia Matki Dziecka i Mlodziezy, Warsaw
  - Centralny Szpital Kliniczny Mswia, Warsaw
  - Reumatika-Centrum Reumatologii, NZOZ, Warsaw
  - NZOZ Vivamed, Warsaw
  - Bodyclinic Sp. z o.o. sp. k, Warsaw
  - Melita Medical Sp. z o.o., Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - Przychodnia Vistamed, Wroclaw
  - EuroMediCare Szpital Specjalistyczny z Przychodnia, Wroclaw
  - Centrum Diagnostyczno - Lecznicze Barska sp. z o.o. Szpital Specjalistyczny Barska, Włocławek
  - ETG Zamosc, Zamość
- Portugal (5):
  - Centro Hospitalar de Lisboa Norte Hospital Santa Maria, Lisbon
  - Uls Loures Odivelas - Hosp. Loures, Loures
  - Hospital de Portimao-Centro Hospitalar do Barlavento Algarvio, Portimão
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E, Santa Maria da Feira
  - Uls Gaia Espinho, Vila Nova de Gaia
- Slovakia (4):
  - FNsP F.D.R. Banska Bystrica, Banská Bystrica
  - Cliniq s.r.o., Bratislava
  - GASTRO I. s.r.o., Prešov
  - Gastroenterology Department ENDOMED, s.r.o., Vranov nad Topľou
- Slovenia (2):
  - Splosna bolnisnica Celje, Celje
  - Univerzitetni klinicni center Ljubljana, Ljubljana
- South Africa (5):
  - Worthwhile Clinical Trials Lakeview Hospital, Benoni
  - Mediclinic Panorama, Cape Town
  - Groote Schur Hospital, Cape Town
  - Practice Dr Naeem Moosa, Johannesburg
  - Emmed Research, Pretoria
- South Korea (14):
  - Inje University Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Chosun university hospital, Gwangju
  - The Catholic university of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea Seoul St.Mary's Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (8):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. La Paz, Madrid
  - Hosp. de Navarra, Pamplona
  - Hosp. Montecelo, Pontevedra
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Univ. de Torrejon, Torrejón de Ardoz
  - Hosp. Alvaro Cunqueiro, Vigo
- Sweden (2):
  - Karolinska Universitetssjukhuset Solna, Solna
  - Ersta sjukhus, Stockholm
- Switzerland (5):
  - Universitatsspital Basel, Basel
  - Inselspital Universitatsspital Bern, Bern
  - Gastroenterologische Praxis Balsiger und Seibold, Bern
  - Kantonsspital St Gallen, Sankt Gallen
  - UniversitaetsSpital Zuerich, Zurich
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Division of Infectious Diseases, Taipei
  - Chang-Gung Memorial Hospital, LinKou Branch, Taoyuan District
- United Kingdom (7):
  - Royal Victoria Hospital, Belfast
  - Addenbrooke's Hospital, Cambridge
  - Queen Elizabeth University Hospital, Glasgow
  - Velocity Clinical Research, High Wycombe
  - Chelsea And Westminster Hospital, London
  - St Georges University Hospital NHS Foundation Trust, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency